CLINICAL TRIAL: NCT00141622
Title: Does Sodium Affect Endothelial Function in Individuals With Chronic Kidney Disease?
Brief Title: Sodium-Endothelial Function-CKD Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: British Heart Foundation (Other); St. George's Hospital Charitable Foundation (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LREC 04/Q0803/181
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2005-08

CONDITIONS: Kidney Failure, Chronic
Keywords: Endothelial dysfunction; ADMA; DDAH; Sodium
MeSH Terms: conditions — Kidney Failure, Chronic

INTERVENTIONS:
Drug: Slow sodium

SUMMARY:
Heart disease and stroke, known as cardiovascular disease, are major causes of death in people with chronic kidney disease. Abnormalities of a metabolic pathway called the "L-arginine-nitric oxide" pathway are thought to be particularly important in these people, and previous research in animals has suggested that sodium (salt) affects part of this metabolic pathway. The purpose of our research is to study the effects of sodium intake on the "L-arginine-nitric oxide" pathway, and on blood vessel function, in patients with kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is associated with abnormalities of endothelial function (EF) and nitric oxide (NO) synthesis, and it is proposed that the endogenous NO synthase inhibitor asymmetrical dimethylarginine (ADMA) plays a central role. In man ADMA is largely metabolized by dimethylarginine dimethylaminohydrolase (DDAH), with some renal excretion occurring. Sodium inhibits DDAH expression in experimental animals and, given that CKD is frequently characterized by sodium retention, it would be interesting to study the effects of sodium loading on DDAH activity/expression, ADMA levels and EF in CKD patients.

To answer these questions, we have designed a double-blind cross-over study employing Slow Sodium (150 mmol/day) and placebo for seven days in individuals with mild-to-moderate CKD. Changes in the ratio of urinary ADMA to dimethylamine (DMA, an ADMA metabolite) will be used as an marker of DDAH activity/expression. ADMA will be measured by ELISA, DMA by high performance liquid chromatography, and EF by venous occlusion plethysmography.

We propose to test the following hypothesis; that in subjects with mild-to-moderate CKD under conditions of high sodium intake, as compared to low-normal sodium intake:

(i) The ratio [ADMA]urine:[DMA]urine is increased (ii) [ADMA]plasma is increased (iii) Endothelium-dependent vasodilatation is reduced

ELIGIBILITY:
Inclusion Criteria:

* CKD Stages 2 and 3 [= calculated creatinine clearance of 30 to 89 ml/min/1.73m2 by Cockcroft-Gault formula]
* 18 to 75 years old

Exclusion Criteria:

* >3 g/24 hours of proteinuria
* Uncontrolled hypertension (systolic BP >160 mmHg, diastolic BP >100 mmHg on/off anti-hypertensive medication)
* Diabetes mellitus
* Tobacco smoking
* Total fasting cholesterol >6 mmol/L
* Uncontrolled heart failure or active IHD
* Chronic liver failure
* Active malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-04; Study Completion 2006-10

PRIMARY OUTCOMES:
Under conditions of high (vs. low sodium intake) ...
(i) The ratio [ADMA]urine:[DMA]urine is increased
(ii) [ADMA]plasma is increased
(iii) Endothelium-dependent vasodilatation is reduced

CONTACTS AND LOCATIONS:
Overall Officials: Timothy WR Doulton, BSc MRCP, Principal Investigator — SGUL
Locations (1):
- Blood Pressure Unit, Department of Cardiac & Vascular Sciences, SGUL, London, United Kingdom